CLINICAL TRIAL: NCT03219437
Title: A Multicenter, Randomized, Double-Blind, Double-Dummy, Active Controlled Study Comparing the Safety and Efficacy of Risankizumab to Methotrexate in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: A Study Comparing the Safety and Efficacy of Risankizumab to Methotrexate in Subjects With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M16-177
Record Dates: First submitted 2017-07-14; First posted 2017-07-17 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Psoriasis
Keywords: ABBV-066; BI 655066
MeSH Terms: conditions — Psoriasis | interventions — risankizumab; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methotrexate (Active Comparator): Participants to receive double-blind methotrexate.
  Interventions: Drug: methotrexate
- Risankizumab (Experimental): Participants to receive double-blind risankizumab.
  Interventions: Drug: risankizumab

INTERVENTIONS:
Drug: risankizumab — subcutaneous (SC) injection
  Other Names: ABBV-066; BI 655066
  Arms: Risankizumab
Drug: methotrexate — capsule
  Arms: Methotrexate

SUMMARY:
The purpose of this study is to compare the safety and efficacy of risankizumab to methotrexate in participants with moderate to severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of plaque psoriasis (with or without concurrent psoriatic arthritis) for at least 6 months before the first administration of study drug
* Have stable moderate to severe plaque psoriasis with or without psoriatic arthritis at both Screening and Baseline Visits
* Be a candidate for systemic therapy for plaque psoriasis as assessed by the investigator
* Be a candidate for treatment with methotrexate (MTX) according to local label

Exclusion Criteria:

* Subjects with non-plaque forms of psoriasis, current drug-induced psoriasis, or active ongoing inflammatory diseases other than psoriasis that might confound study evaluations according to investigator's judgment
* Previous exposure to risankizumab
* Previous exposure to MTX
* Use of any prohibited medication or any drug considered likely to interfere with the safe conduct of the study, as assessed by the investigator
* Subject has a history of clinically significant hematologic, renal, or liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2021-11-26 (Actual); Study Completion 2021-11-26 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with Static Physician Global Assessment (sPGA) score of clear or almost clear (0, 1) at Week 28. | Week 28
  The sPGA is the physician's current assessment of the average thickness, erythema, and scaling of all psoriatic lesions.
Percentage of participants with a ≥ 90% reduction from Baseline Psoriasis Area and Severity Index (PASI 90) at Week 28 | Week 28
  PASI90 denotes greater than or equal to 90% improvement in PASI score. PASI provides a quantitative assessment of psoriasis disease state based on the amount of body surface area that is affected and the degree of severity of erythema, induration, and scale, weighted by body part.

SECONDARY OUTCOMES:
Percentage of participants with a 100% reduction from Baseline PASI score (PASI 100) at Week 28 | Week 28
  PASI100 denotes greater than or equal to 100% improvement in PASI score. PASI provides a quantitative assessment of psoriasis disease state based on the amount of body surface area that is affected and the degree of severity of erythema, induration, and scale, weighted by body part.
Percentage of participants with a ≥ 75% reduction from Baseline PASI score (PASI 75) at Week 28 | Week 28
  PASI75 denotes greater than or equal to 75% improvement in PASI score. PASI provides a quantitative assessment of psoriasis disease state based on the amount of body surface area that is affected and the degree of severity of erythema, induration, and scale, weighted by body part.
Percentage of participants with Static Physician Global Assessment (sPGA) score of clear (0) at Week 28 | Week 28
  The sPGA is the physician's current assessment of the average thickness, erythema, and scaling of all psoriatic lesions.
Change from baseline in EQ-5D-5L at all visits collected | Week 28
  The EQ-5D-5L is a standardized non-disease specific instrument for describing and valuing health-related quality of life.
Achievement of an increase of 0.1 or more points from baseline in European Quality of Life 5 Dimensions (EQ-5D-5L) at all visits | Week 28
  The EQ-5D-5L has five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. These dimensions are measured on a five-level scale: no problems, slight problems, moderate problems, severe problems, and extreme problems.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (11):
- Brazil (11):
  - CETI - Centro de Estudos em Terapias Inovadoras /ID# 208593, Curitiba, Paraná
  - PUC Trials-Nucleo de Pesquisa clinica da Escola de Medicina da PUCPR /ID# 164401, Curitiba, Paraná
  - Hospital Moinhos de Vento /ID# 208592, Porto Alegre, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre /ID# 164565, Porto Alegre, Rio Grande do Sul
  - Unidade de Pesquisa Clínica da Faculdade de Medicina de Botucatu /ID# 164743, Botucatu, São Paulo
  - Hospital de Clinicas da Universidade Estadual de Campinas - UNICAMP /ID# 164521, Campinas, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto - USP /ID# 164768, Ribeirão Preto, São Paulo
  - Faculdade de Medicina do ABC /ID# 164519, Santo André, São Paulo
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto /ID# 164723, São José do Rio Preto, São Paulo
  - Instituto de Dermatologia e Estética do Brasil /ID# 164754, Rio de Janeiro
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo /ID# 164805, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=M16-177&Latitude=&Longitude=&LocationName=#additional-resources-section